CLINICAL TRIAL: NCT01879839
Title: Phase 4 Study of Effect of a Pre-interventional Calorie Restriction on Renal Function After Administration of Contrast Agent in Patients at Risk
Brief Title: Effect of a Pre-interventional Diet on Renal Function After Administration of Contrast Agent in Patients at Risk
Acronym: CR_KMN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, MD, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: uni-koeln-1547; 2012-003696-18 (EudraCT Number)
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Renal Failure Chronic Contrast Induced
MeSH Terms: interventions — Diet

STUDY DESIGN:
Intervention Model Description: One arm with controlled diet, second arm as control group with no diet.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Patients who don't follow a special diet.
- Diet Group (Other): Patients who subsist on a special diet.
  Interventions: Dietary Supplement: Diet

INTERVENTIONS:
Dietary Supplement: Diet — Patients receive special diet 4 days prior to contrast-agent administration.
  Arms: Diet Group

SUMMARY:
The aim of this study is to assess the effect of a diet prior to administration of contrast agent in terms of a preventive procedure which leads to an attenuation of the contrast-induced nephropathy (CIN).

Patients with a known kidney disease are especially at risk. A potential beneficial effect of a diet prior to intervention has been shown in investigations in mammals, therefore this study will investigate if a pre-interventional diet in patients with known kidney disease and scheduled contrast agent examination can attenuate or prevent a post-interventional loss of kidney function.

DETAILED DESCRIPTION:
Patients with contrast agent examinations are at risk for contrast-induced nephropathy (CIN) and in succession acute renal failure which is associated with significant morbidity and mortality. None of the currently used preventive procedures show a benefit in terms of a CIN-prevention.

Experimental data suggests, that a pre-interventional caloric restriction might provide kidney protection in this context. This clinical trial investigates if this phenomenon is also applicable in humans. Patients with increased risk for a post-interventional renal failure due to known chronic kidney disease are randomized in 2 groups. Patients of the diet group receive a calorie restriction to 60% of the calculated daily energy rate from day -4 until day -1 (included) pre-intervention (day 0 corresponds to day of intervention). Patients of the control group receive alimentation ad libitum.

Primary objective is the increase of serum creatinine in mg/dl 48 h after begin of intervention in comparison to baseline value obtained in the morning of the day of intervention (day 0) in order to analyse if a pre-interventional calorie restriction as a preventive strategy leads to an attenuation of post-interventioal kidney injury.

Hypothesis: A four day calorie restriction reduces the increase of serum creatinine after administration of contrast agent in patients with known chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. men and women 18 years of age or older
2. caucasian origin
3. scheduled coronary angiography
4. indication for coronary angiography is determined by the referring physician
5. Patient and/or legal guardian must be willing and able to give written informed consent
6. at least one of the following risk factors:

   * serum creatinine > 1,1 mg/dl in male patients or serum creatinin > 0,9 mg/dl in female patients
   * Type 2 diabetes
   * peripher arteriovascular disease
   * heartfailure with NYHA 3-4 or ejection fraction ≤ 50%
   * age over 70 years

Exclusion Criteria:

1. End-stage renal disease (patient on dialysis)
2. Indwelling kidney transplant
3. Malnutrition (BMI < 18,5 kg/m2)
4. Body weight < 46 kg in male, < 51 kg in female
5. BMI > 35 kg/m2 or body weight > 120 kg
6. diet within the previous 4 weeks
7. Inappetence
8. Weight loss > 1 kg within the previous 2 weeks, if not explained by use of diuretics
9. Consuming underlying disease 10. Uncontrolled local or systemic infection 11. Contraindication for enteral nutrition 12. Known allergy against or incompatibility with ingredients of the employed formula-diet 13. Pregnancy or breast feeding 14. Participation in other interventional clinical trials 15. Missing safe method of contraception or missing occurence of menopause (in female) 16. Professional or private relationship between subject and the investigators or dependence on the investigators 17. Placement in an institution based on official orders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Rise of serum creatinine in mg/dl 48 hours after begin of coronary intervention (contrast agent administration) | Baseline to 48 hours

SECONDARY OUTCOMES:
Rise of serum creatinine in mg/dl 24 hours after begin of coronary intervention. | Baseline to 24 hours
Neutrophile-Gelatinase associated Lipocaline (NGAL in µg/l) in urine 24 hours after begin of coronary intervention. | Baseline to 24 hours
Cystatin C in Plasma (mg/l) 24 hours after begin of coronary intervention. | Baseline to 24 hours

OTHER OUTCOMES:
Occurrence of CIN (contrast-agent induced nephropathy) with rise of serum creatinine about ≥ 0,5 mg/dl or ≥ 25% of initial value with 48 hours. | Baseline to 48 hours.
Occurrence of acute renal failure corresponding KDIGO I, II, III | Baseline to 4 weeks
Necessity of dialysis up to 4 weeks after coronary intervention. | Baseline to 4 weeks.
Mortality at timepoint 4 weeks after coronary intervention. | Baseline to 4 weeks.
Hospitalization up to 4 weeks after coronary intervention. | Baseline to 4 weeks.
Urea (mg/dl), white blood cells (/µl) LDH (U/l), CRP (mg/l), CK (U/l), CK-MB (U/l und %) at timepoint 24 and 48 hours after coronary angiography | Baseline to 24 and 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Principal Investigator — University of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Germany